CLINICAL TRIAL: NCT07290608
Title: Clinical Performance of the DOACT Algorithm Versus AI-Based Decision Models in Oral Anticoagulant Therapy for Vascular Patients
Brief Title: DOACT Algorithm Versus AI-Based Decision Models in Oral Anticoagulant Therapy for Vascular Patients
Acronym: DOACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ITALO EUGENIO SOUZA GADELHA DE ABREU (Other)
Responsible Party: Sponsor-Investigator, ITALO EUGENIO SOUZA GADELHA DE ABREU, Principal Investigator, Science Valley Research Institute
Organization: Science Valley Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DOACT-AI-VASC Study
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Deep Vein Thrombosis; Superficial Thrombophlebitis; Pulmonary Thromboembolisms; Clinical Decision Support Systems; Artificial Intelligence
Keywords: anticoagulant; algorithm; thrombosis
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Intervention Model Description: Three-arm comparative validation study evaluating the accuracy and clinical utility of the DOACT algorithm versus standard clinical decision-making and large language model (LLM)-based decision tools.
Who Masked: Investigator
Masking Description: Single-blind. Investigator was blinded to the intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DOACT algorithm (Experimental): Use of DOACT algorithm (Dose-Oriented Anticoagulant Calculator for Evidence-Based Decision Tool) to recommend appropriate oral anticoagulant regimens.
  Interventions: Other: DOACT algorithm
- No algorithm (Placebo Comparator): Standard clinical decision-making to recommend appropriate oral anticoagulant regimens.
  Interventions: Other: No algorithm
- LLM-based tools (Active Comparator): Use of large language model (LLM)-based tools to recommend appropriate oral anticoagulant regimens.
  Interventions: Other: LLM-based tools

INTERVENTIONS:
Other: DOACT algorithm — Vascular and non-vascular physicians using DOACT (Dose-Oriented Anticoagulant Calculator for Evidence-Based Decision Tool) to recommend appropriate oral anticoagulant regimens-dose selection and duration responding 15 standardized clinical case vignettes representing patients with vascular diseases such as deep vein thrombosis (DVT), superficial thrombophlebitis, and pulmonary thromboembolism (PTE).
  Arms: DOACT algorithm
Other: No algorithm — Vascular and non-vascular physicians using standard clinical decision-making (no use of algorithm) to recommend appropriate oral anticoagulant regimens-dose selection and duration responding 15 standardized clinical case vignettes representing patients with vascular diseases such as deep vein thrombosis (DVT), superficial thrombophlebitis, and pulmonary thromboembolism (PTE).
  Arms: No algorithm
Other: LLM-based tools — Vascular and non-vascular physicians using large language model (LLM)-based tools to recommend appropriate oral anticoagulant regimens-dose selection and duration responding 15 standardized clinical case vignettes representing patients with vascular diseases such as deep vein thrombosis (DVT), superficial thrombophlebitis, and pulmonary thromboembolism (PTE).
  Arms: LLM-based tools

SUMMARY:
Study using a decision algorithm for the application of an oral anticoagulant calculator in vascular diseases, aimed at validating a clinical decision-support tool for conditions such as deep vein thrombosis, superficial thrombophlebitis, and pulmonary thromboembolism.

DETAILED DESCRIPTION:
Cross-sectional, three-arm comparative validation study evaluating the accuracy and clinical utility of the DOACT algorithm versus standard clinical decision-making and large language model (LLM)-based decision tools.

ELIGIBILITY:
Inclusion Criteria

* Physicians with residency training in Vascular Surgery or official Board Certification in Vascular Surgery.
* Currently practicing clinical and/or surgical vascular care in Brazil.
* Completed the informed consent process (TCLE) and voluntarily agreed to participate.

Exclusion Criteria

* Physicians without formal Vascular Surgery residency and without Board Certification.
* Physicians not performing vascular clinical or surgical care (e.g., exclusively administrative, academic, or non-assistance roles).
* Less than 1 year of professional experience after medical school graduation.
* Did not sign or did not fully complete the TCLE.

Large Language Models (LLMs)

* Inclusion Criteria
* Free-access LLMs available to the public at the time of data collection.
* All responses generated using the same standardized prompt.
* Capable of producing complete, text-based clinical answers relevant to vascular surgery decision-making.

Exclusion Criteria

* Paid or subscription-based LLMs.
* LLMs requiring institutional licenses, restricted access, or proprietary tokens.
* Models unable to generate full responses to the standardized prompt.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of the DOACT Algorithm in Guiding Oral Anticoagulant Therapy | Day 1
  Accuracy of anticoagulation recommendations
  Description: Proportion of correct responses generated by the four evaluated LLMs, vascular surgeons, and non-vascular physicians, with and without access to the DOACT algorithm, using standardized clinical vignettes.
Accuracy of anticoagulation recommendations | Day 1
  Proportion of correct responses generated by LLMs, vascular surgeons, and non-vascular physicians with and without access to the DOACT algorithm. All LLM outputs will be generated using the same standardized prompt, following methodological guidance recommended by IBM for evaluating large language models.

OTHER OUTCOMES:
1. Identification of key clinical elements 2.Response time | Day 1
  Correct reporting of dosing adjustments, renal criteria, bleeding risks, reversal agents, and contraindications.
  Description: Time (seconds) from prompt submission to full answer generation for LLMs, and time to completion for physicians.

CONTACTS AND LOCATIONS:
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gee E. The National VTE Exemplar Centres Network response to implementation of updated NICE guidance: venous thromboembolism in over 16s: reducing the risk of hospital-acquired deep vein thrombosis or pulmonary embolism (NG89). Br J Haematol. 2019 Sep;186(5):792-793. doi: 10.1111/bjh.16010. Epub 2019 Jun 5. No abstract available. PMID 31168834
- [Background] Vinogradova Y, Coupland C, Hill T, Hippisley-Cox J. Risks and benefits of direct oral anticoagulants versus warfarin in a real world setting: cohort study in primary care. BMJ. 2018 Jul 4;362:k2505. doi: 10.1136/bmj.k2505. PMID 29973392
- [Background] Nielsen PB, Lundbye-Christensen S, Rasmussen LH, Larsen TB. Improvement of anticoagulant treatment using a dynamic decision support algorithm: a Danish Cohort study. Thromb Res. 2014 Mar;133(3):375-9. doi: 10.1016/j.thromres.2013.12.042. Epub 2014 Jan 7. PMID 24444650
- [Background] Kakkos SK, Gohel M, Baekgaard N, Bauersachs R, Bellmunt-Montoya S, Black SA, Ten Cate-Hoek AJ, Elalamy I, Enzmann FK, Geroulakos G, Gottsater A, Hunt BJ, Mansilha A, Nicolaides AN, Sandset PM, Stansby G, Esvs Guidelines Committee, de Borst GJ, Bastos Goncalves F, Chakfe N, Hinchliffe R, Kolh P, Koncar I, Lindholt JS, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, De Maeseneer MG, Comerota AJ, Gloviczki P, Kruip MJHA, Monreal M, Prandoni P, Vega de Ceniga M. Editor's Choice - European Society for Vascular Surgery (ESVS) 2021 Clinical Practice Guidelines on the Management of Venous Thrombosis. Eur J Vasc Endovasc Surg. 2021 Jan;61(1):9-82. doi: 10.1016/j.ejvs.2020.09.023. Epub 2020 Dec 15. No abstract available. PMID 33334670